CLINICAL TRIAL: NCT03709602
Title: Social Determinants of HPV Vaccine Completion Among Adolescents
Brief Title: SDH of HPV Vaccine Completion
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00100733
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Results first posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Human Papilloma Virus
Keywords: HPV; adolescents; HPV Vaccine; social determinants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adolescents ages 11 to 14 years: Adolescents ages 11 to 14 years who have received 1 dose of the HPV vaccine series between January 2017 and December 2017
- Parent of adolescents: Parents as defined as the adolescent's biological mother or father, step-parents, or legal guardian, and who self-identified as the primary caregiver of the adolescent child and most likely to make medical decisions for the adolescent.
- Cohort of Adolescents From Electronic Health Record (EHR): A cohort of adolescents ages 11 to 14 who received 1 dose of the HPV vaccine from January 2017 to December 2017 within the university's health system network. The cohort was followed from January 2018 to February 2019 to assess vaccine completion within a 14-month period.

SUMMARY:
The purpose of this research study is to find out which factors influence parents' ability to complete the human papillomavirus (HPV) vaccine series for their child. The information learned from this study may help the investigators develop programs to improve HPV vaccine completion rates among adolescents and reduce barriers to receiving the second shot of the vaccine series.

ELIGIBILITY:
Inclusion Criteria:

* For adolescents, participants need to be between the ages 11 to 14 years.
* Received 1 dose of the HPV vaccine series between January 2017 and December 2017.
* For parents, there is no age limit required.
* Parents as defined as the adolescent's biological mother or father, step-parents, or legal guardian.
* Parents or legal guardians who self-identified as the primary caregiver of the adolescent child and most likely to make medical decisions for the adolescent.

Exclusion Criteria:

* Parents with cognitive impairment.
* Adolescents with cognitive impairment.
* Adolescents emancipated from their parents or legal guardian
* Pregnant adolescent girls.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Adolescents ages 11 to 14 years and their parent from Duke University Primary Care Pediatrics at Roxboro Road.
Sampling Method: Non-Probability Sample
Enrollment: 3076 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Gonzalez-Guarda, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Primary Care Pediatrics at Roxboro Road, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 32 participants were recruited for the qualitative portion of the study to participate in interviews (n = 16 parents, n = 16 adolescents)
Pre-assignment Details: Cohort of Adolescents from electronic health record group were reviewed retrospectively from January 1, 2017- February 28, 2019. Enrollment of parents and adolescents (n = 32) began on the start date of January 7, 2019.
Groups:
- Adolescents Ages 11 to 14 Years: Adolescents ages 11 to 14 years who have received 1 dose of the HPV vaccine series between January 2017 and December 2017. Adolescents were stratified into two groups: Completer (defined as adolescents who received two vaccine doses within a 14-month period) and Non-Completer (defined as adolescents who received only one vaccine dose within 14-month period). Qualitative sample.
- Parent of Adolescents: Parents as defined as the adolescent's biological mother or father, step-parents, or legal guardian, and who self-identified as the primary caregiver of the adolescent child and most likely to make medical decisions for the adolescent. Parents were stratified into two groups (Completer or Non-Completer as described in the adolescent group) based on the adolescent's vaccination status. Qualitative sample.
- Cohort of Adolescents From Electronic Health Record (EHR): A cohort of adolescents ages 11 to 14 who received 1 dose of the HPV vaccine from January 2017 to December 2017 within the university's health system network. The cohort was followed from January 2018 to February 2019 to assess vaccine completion within a 14-month period. Quantitative sample.
Period: Overall Study
Arm/Group | Adolescents Ages 11 to 14 Years | Parent of Adolescents | Cohort of Adolescents From Electronic Health Record (EHR)
Started | 16 (Adolescents recruited for qualitative interviews.) | 16 (Parents recruited for qualitative interviews.) | 3044 (Cohort of adolescents created from the EHR data for the quantitative portion of the study.)
Completed | 16 (Adolescents recruited for qualitative interviews.) | 16 (Parents recruited for qualitative interviews.) | 3044 (Cohort of adolescents created from the EHR data for the quantitative portion of the study.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: There is no quantitative results beyond demographics for the Adolescents ages 11 to 14 years and parent of adolescents groups as this was not part of the aim of the study.
Groups:
- Adolescents Ages 11 to 14 Years: Adolescents ages 11 to 14 years who have received 1 dose of the HPV vaccine series between January 2017 and December 2017. Adolescents were stratified into two groups: Completer (defined as adolescents who received two vaccine doses within a 14-month period) and Non-Completer (defined as adolescents who did not receive two vaccine doses). Qualitative sample.
- Total: Total of all reporting groups
Arm/Group | Adolescents Ages 11 to 14 Years | Parent of Adolescents | Cohort of Adolescents From Electronic Health Record (EHR) | Total
Number analyzed (Participants) | 16 | 16 | 3044 | 3076
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 0 | 3044 | 3060
  Between 18 and 65 years | 0 | 16 | 0 | 16
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 12 [11 to 14] | 43 [29 to 67] | 12.1 [11 to 14] | NA [NA to NA] — The mean age for the participant sample of parents for the qualitative interviews were analyzed separately from the cohort of adolescent group using the EHR dataset, since parents were not included in the quantitative dataset.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 16 | 1492 | 1517
  Male | 7 | 0 | 1552 | 1559
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 215 | 225
  Not Hispanic or Latino | 11 | 11 | 2653 | 2675
  Unknown or Not Reported | 0 | 0 | 176 | 176
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The sample size of the cohort of adolescent group for the race variable differs from overall quantitative sample population (N=3044) because race information was not provided for some participants who reported Hispanic ethnicity.
  Participants
    American Indian or Alaska Native | 0 | 0 | 12 | 12
    Asian | 0 | 0 | 118 | 118
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 2
    Non Hispanic Black or African American | 6 | 5 | 965 | 976
    Non-Hispanic White | 3 | 5 | 1441 | 1449
    More than one race | 2 | 1 | 82 | 85
    Hispanic Other | 4 | 4 | 131 | 139
    Hispanic White | 1 | 1 | 0 | 2
    Non-Hispanic Other | 0 | 0 | 33 | 33
    Unknown or Not Reported | 0 | 0 | 176 | 176
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 16 | 3044 | 3076
HPV vaccine completion status [Count of Participants; unit: Participants] — Completer defined as receiving 2 or 3 vaccine doses within 14-month period determined by the CDC's vaccine administration schedule. Non-completer defined as receiving only 1 vaccine dose within 14-month period.
  Participants
    Completers | 8 | 8 | 1961 | 1977
    Non-Completers | 8 | 8 | 1083 | 1099

OUTCOME MEASURES:

1. Primary Outcome: Overall HPV Vaccine Completion Rates
Description: Adolescents who completed the required HPV vaccine doses (e.g. two or three doses based on the CDC's vaccine administration guidelines for adolescents' ages 11 to 14 years) during the January 2017 to February 2019 observation period.
Time Frame: up to 14 months
Population: Vaccine completion rates were only analyzed for the quantitative sample of adolescents using the EHR data (N=3044).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort of Adolescents From Electronic Health Record (EHR)
Number analyzed (Participants) | 3044
Participants
  Completers | 1961
  Non-Completers | 1083

2. Secondary Outcome: HPV Vaccine Completion Within 14-Months
Description: Adolescents who received the required number of doses for vaccine completion, defined as the receipt of two or three doses based on the CDC's guidelines for adolescents' ages 11 to 14 years, within 14-months from their first vaccine dose.
Time Frame: within 14 months
Population: Vaccine completion rates were only analyzed for the quantitative sample of adolescents using the EHR data (N=3044).
Measure: Count of Participants; unit: Participants
Groups:
- Cohort of Adolescents From EHR: A cohort of adolescents ages 11 to 14 who received 1 dose of the HPV vaccine from January 2017 to December 2017 within the university's health system network. The cohort was followed from January 2018 to February 2019 to assess vaccine completion within a 14-month period.
Arm/Group | Cohort of Adolescents From EHR
Number analyzed (Participants) | 3044
Participants | 1637

ADVERSE EVENTS:
Time Frame: 1 year
Description: Participants in the Cohort of Adolescents From EHR group were not monitored/assessed for adverse events.
Groups:
- Adolescents Ages 11 to 14 Years: Adolescents ages 11 to 14 years who have received 1 dose of the HPV vaccine series between January 2017 and December 2017. Adolescents were stratified into two groups: Completer (defined as adolescents who received two vaccine doses within a 14-month period) and Non-Completer (defined as adolescents who did not receive two vaccine doses).
- Parent of Adolescents: Parents as defined as the adolescent's biological mother or father, step-parents, or legal guardian, and who self-identified as the primary caregiver of the adolescent child and most likely to make medical decisions for the adolescent. Parents were stratified into two groups (Completer or Non-Completer as described in the adolescent group) based on the adolescent's vaccination status.
Arm/Group | Adolescents Ages 11 to 14 Years | Parent of Adolescents
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT03709602/Prot_SAP_000.pdf